CLINICAL TRIAL: NCT05584384
Title: The Application of New Diagnostic (Thermovision) and Treatment (tDCS) Procedures in Patients With Drug-resistant Orofacial Pain
Brief Title: The Use of tDCS in the Orofacial Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Tadeáš Mareš, Head of tDCS lab, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 53/22 Grant AZV VES 2023VFN
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Orofacial Pain
Keywords: Orofacial Pain; tDCS; trancranial DIrect Current Stimulation; NIBS; non-invasive brain stimulation
MeSH Terms: conditions — Facial Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blinded, placebo-controlled, two-arm trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants will be distributed between 2 arms using an aperiodic, nondeterministic, atmospheric random noise randomization algorithm. The stimulation type will be unblinded upon completing all the follow-ups or dropping out. The blinding will be ensured by a dedicated team member with no direct access to the participants or their data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): The investigators aim for six sessions of anodal stimulation over the right primary motor area contralateral to the orofacial pain (C3 or C4 in 10-20 EEG system) with cathode above the frontal area ipsilateral to the orofacial pain (Fp1 or Fp2) using HDCstim by Newronika S.r.l., Italy. The therapy will be administered over two weeks (Mon, Wed, Fri) to ensure a washout period of 48 to 72 hours between applications. The current of 2 mA will be delivered via silicone electrodes inserted into saline (0.9%) filled cellulose sponges, anode 5x5cm, cathode 6x8cm, for 20 minutes with 20 seconds of both ramp-up and ramp-down. An International 10-20 EEG system will be used to determine the stimulation location, and dedicated EEG caps will be used to ensure consistency between applications.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham group (Placebo Comparator): The sham (placebo) will be administered using the same devices with a preprogrammed sham protocol (using HDCprog by Newronika S.r.l., Italy) of 20 minutes to be virtually indistinguishable from the active stimulation.
  Interventions: Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial Direct Current Stimulation (tDCS) is a non-invasive neuromodulatory method utilizing weak electrical currents to elicit short and long-term central nervous system changes.
  Other Names: tDCS
  Arms: Active group
Device: Sham Transcranial Direct Current Stimulation — The sham was administered using the same tDCS devices as in the active group with a preprogrammed sham protocol of 20 minutes to be virtually indistinguishable from the active stimulation.
  Other Names: Sham tDCS
  Arms: Sham group

SUMMARY:
The trial´s main goal is to explore the use of transcranial direct current stimulation (tDCS) as a treatment option for persons suffering from orofacial pain. The aim of the trial is to further investigate the efficacy and longevity of tDCS in treating chronic pharmacoresistant orofacial pain.

A prospective, randomized, double-blinded, two-arm, sham-controlled design will be utilized. Primarily, the analgesic effect's intensity and duration will be assessed. Secondarily, the associated reduction of symptoms of anxiety and depression will be investigated, as well as the impact on the general quality of life. Anodal stimulation (6 sessions in 2 weeks, 2mA, 20 min, cathode over the opposite Fp area) of M1 contralateral to the pain location will be employed. Washout periods of 48-72 hours will be kept between applications to improve neuroplasticity changes' induction, which is estimated to reflect in the effect retention. Eight major evaluation points will be employed in 26 weeks, and a daily numeric rating scale (NRS) self-assessment.

The trial will potentially improve the quality of life, reduce the health burden caused by chronic orofacial pain, and provide further data on the use of tDCS in this setting, thus, enabling an additional route to manage the symptoms of pain in the future.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Orofacial Pain by a pain medicine specialist according to ICOP (International classification of orofacial pain) and ICHD3 (International classification of headache disorder)
* Stable analgesic therapy one month before the stimulation series

Exclusion Criteria:

* Changes to the analgesic therapy in 6 months following the stimulation series
* Non-compliance with the follow-ups
* General contraindications to tDCS - pregnancy, unstable cardiovascular disorders, epilepsy and intracranial masses

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The McGill Pain Questionnaire (short form). | The measurement will be established as a baseline prior to the stimulation series. (at T1)
  The Short-form McGill Pain Questionnaire is a standardized questionnaire assessing pain's sensory and affective dimensions. The types of pain are scaled as to their intensity between 1-4 (a higher value denotes higher intensity), the overall intensity is scaled between 0-5 (a higher value denotes higher intensity), and VAS is used to visualize the notion of pain (evaluated on a scale of 0-10, a higher value denotes higher intensity).
Changes in The McGill Pain Questionnaire (short form) at T2. | Measured at T2 (after the 6th stimulation, 2 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in The McGill Pain Questionnaire (short form) at T3. | Measured at T3 (6 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in The McGill Pain Questionnaire (short form) at T4. | Measured at T4 (10 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in The McGill Pain Questionnaire (short form) at T5. | Measured at T5 (14 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in The McGill Pain Questionnaire (short form) at T6. | Measured at T6 (18 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in The McGill Pain Questionnaire (short form) at T7. | Measured at T7 (22 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in The McGill Pain Questionnaire (short form) at T8. | Measured at T8 (26 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
The numeric rating scale (NRS) as part of "pain diary" | The measurement will be established as a baseline prior to the stimulation series. (at T1)
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable.
Changes in the numeric rating scale (NRS) every day of them follow-up period. | Measured every day since T1 up until T8. (for 26 weeks in total)
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable.
The Margolis Pain Diagram | The measurement will be established as a baseline prior to the stimulation series. (at T1)
  The Margolis pain diagram weights the extension and distribution of pain, expressed as the percentage of body surface in pain and its location. The tool consists of a dorsal and a ventral drawing of the body. The subjects are asked to shade areas in which they have experienced pain.
Changes in the Margolis Pain Diagram at T2. | Measured at T2 (after the 6th stimulation, 2 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in the Margolis Pain Diagram at T3. | Measured at T3 (6 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in the Margolis Pain Diagram at T4. | Measured at T4 (10 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in the Margolis Pain Diagram at T5. | Measured at T5 (14 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in the Margolis Pain Diagram at T6. | Measured at T6 (18 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in the Margolis Pain Diagram at T7. | Measured at T7 (22 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in the Margolis Pain Diagram at T8. | Measured at T8 (26 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
The questionnaire of interference with daily activities | The measurement will be established as a baseline prior to the stimulation series. (at T1)
  A standardized questionnaire to evaluate the interference of pain with daily activities. Minimum=0 points, maximum=5 points. A higher score generally means more severe interference.
Changes in the questionnaire of interference with daily activities at T2. | Measured at T2 (after the 6th stimulation, 2 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in the questionnaire of interference with daily activities at T3. | Measured at T3 (6 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in the questionnaire of interference with daily activities at T4. | Measured at T4 (10 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in the questionnaire of interference with daily activities at T5. | Measured at T5 (14 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in the questionnaire of interference with daily activities at T6. | Measured at T6 (18 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in the questionnaire of interference with daily activities at T7. | Measured at T7 (22 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in the questionnaire of interference with daily activities at T8. | Measured at T8 (26 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement

SECONDARY OUTCOMES:
Beck's Depression Inventory (BDI) | The measurement will be established as a baseline prior to the stimulation series. (at T1)
  A standardized questionnaire to evaluate the symptoms of depression. Minimum=0 points, maximum=63 points. A higher score generally means more severe anxiety
Changes in Beck's Depression Inventory (BDI) at T2. | Measured at T2 (after the 6th stimulation, 2 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in Beck's Depression Inventory (BDI) at T3. | Measured at T3 (6 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in Beck's Depression Inventory (BDI) at T4. | Measured at T4 (10 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in Beck's Depression Inventory (BDI) at T5. | Measured at T5 (14 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in Beck's Depression Inventory (BDI) at T6. | Measured at T6 (18 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in Beck's Depression Inventory (BDI) at T7. | Measured at T7 (22 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in Beck's Depression Inventory (BDI) at T8. | Measured at T8 (26 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Beck Anxiety Inventory (BAI) | The measurement will be established as a baseline prior to the stimulation series. (at T1)
  A standardized questionnaire to evaluate the symptoms of anxiety. Minimum=0 points, maximum=63 points. A higher score generally means more severe anxiety
Changes in Beck Anxiety Inventory (BAI) at T2. | Measured at T2 (after the 6th stimulation, 2 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in Beck Anxiety Inventory (BAI) at T3. | Measured at T3 (6 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in Beck Anxiety Inventory (BAI) at T4. | Measured at T4 (10 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in Beck Anxiety Inventory (BAI) at T5. | Measured at T5 (14 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in Beck Anxiety Inventory (BAI) at T6. | Measured at T6 (18 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in Beck Anxiety Inventory (BAI) at T7. | Measured at T7 (22 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement
Changes in Beck Anxiety Inventory (BAI) at T8. | Measured at T8 (26 weeks since T1)
  Changes compared to the baseline (T1) will be calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement

CONTACTS AND LOCATIONS:
Overall Officials: Jitka Fricova, M.D., Ph.D., Study Director — General University Hospital in Prague; Charles University in Prague; Tadeas Mares, M.D., Study Chair — General University Hospital in Prague; Charles University in Prague; Martin Anders, M.D., Ph.D., Study Chair — General University Hospital in Prague; Charles University in Prague; Jozef Buday, M.D., Ph.D., Study Chair — General University Hospital in Prague; Charles University in Prague
Locations (1):
- Pain Management Centre, General University Hospital in Prague; Charles University in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
IPD is to be shared on request by a verified researcher. The study director´s discretion is reserved.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When the results are published, indefinitely.
Access Criteria: Verified researchers only.